CLINICAL TRIAL: NCT01898013
Title: Neurosteroids as Novel Therapeutic Agents for Chronic Pain in OEF/OIF Veterans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01710; 1IK2RX000908-01A1 (NIH)
Record Dates: First submitted 2013-07-08; First posted 2013-07-12 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Lower Back Pain
Keywords: pain; pregnenolone; Veterans; clinical trial; neurosteroid; allopregnanolone; low back; placebo controlled; randomized; musculoskeletal
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Pregnenolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregnenolone (Active Comparator): Pregnenolone fixed escalating up to 500mg/day will consist of the following schedule:
  Visit 1 (week -1, screening visit) and pain symptom assessment (no study medication) Visit 2 (week 0) placebo lead-in (all participants) Visit 3 (week 1, baseline visit): 50mg PO, BID x 1 week, Visit 4 (week 2): 150mg PO, BID x 1 week, Visit 5 (week 3): 250mg PO, BID for two weeks. Visit 6 (week 5): No medication will be dispensed; study medication will be tapered by 100mg per day and then discontinued.
  Interventions: Drug: Pregnenolone
- Placebo (Placebo Comparator): Placebo will be administered exactly the same as the active comparator (pregnenolone) and will consist of the following schedule:
  Visit 1 (week -1, screening visit) and pain symptom assessment (no study medication) Visit 2 (week 0) placebo lead-in (all participants) Visit 3 (week 1, baseline visit): placebo PO, BID x 1 week, Visit 4 (week 2): placebo PO, BID x 1 week, Visit 5 (week 3): placebo PO, BID for two weeks. Visit 6 (week 5): No medication will be dispensed; study medication will be tapered in the exact manner as active study medication and then discontinued.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregnenolone
  Arms: Pregnenolone
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study design is a randomized, double-blind, two-arm trial of pregnenolone and placebo to determine the possible analgesic effects in OEF/OIF Veterans with chronic low back pain. The total study duration is 6 weeks (followed by two-follow up phone calls). All patients will monitor pain symptoms for one week with pain diaries, followed by a 1-week placebo-only lead-in period, 90 subjects will be randomly assigned to one of two groups. Of these subjects, 45 subjects will receive pregnenolone, and 45 subjects will receive placebo for 4 weeks. Patient interview assessments and laboratory studies will be performed at each interview time point. Pregnenolone, allopregnanolone and other neurosteroid metabolites will be determined by gas chromatography / mass spectrometry (GC/MS), proceeded by high performance liquid chromatography (HPLC).

ELIGIBILITY:
Inclusion Criteria:

1. OEF/OIF Veterans, 18-65 years of age, with chronic low back pain.
2. Based on medical history and medical records, have low back pain (Thoracic Vertebrae 6 or below) present on most days for the preceding 6 months or longer, and fulfill all disease diagnostic criteria (please see disease diagnostic criteria below).
3. Have a weekly mean of 24-hour average pain score ≥ 4 at baseline.
4. Negative pregnancy test if female. Sexually active subjects are required to use a medically acceptable form of birth control if they are of childbearing potential and could become pregnant during the study. A medically acceptable form of birth control includes non-hormonal intrauterine devices, surgical sterilization, or double barrier methods (e.g., diaphragm with contraceptive jelly, condom with contraceptive foam, cervical caps with contraceptive jelly). Sexual abstinence with agreement to continue abstinence or to use a medically acceptable method of contraception (as listed above) should sexual activity occur is permissible.
5. No change in medications less than 4 weeks before baseline.
6. No anticipated need to alter psychotropic or pain medications for the 6-wk study duration (as determined by study physician's review of records and/or discussion with prescribing physician).
7. Ability to fully participate in the informed consent process.

Exclusion Criteria:

1. Unstable medical or neurological illness, including seizures, renal impairment or cerebral vascular accident.
2. Use of oral contraceptives or other hormonal supplements.
3. Significant suicidal or homicidal ideation requiring intervention.
4. Daily use of long or short-acting narcotic medications.
5. Current Diagnostic and Statistical Manual (DSM-IV) diagnosis of bipolar disorder, schizophrenia, or other psychotic disorder, or cognitive disorder due to a general medical condition (other than if related to mild TBI).
6. Female patients who are pregnant or breast-feeding.
7. Known allergy to study medication.
8. History of moderate or severe TBI (mild TBI is permissible).
9. DSM-IV criteria met for alcohol and/or other substance abuse or dependence within past three months (excludes caffeine and nicotine).
10. Have received epidural steroids, facet block, nerve block, or other invasive procedures aimed to reduce low back pain within the past 3 months prior to Visit 1.
11. Completion of daily diaries for less than 70% of days between Visit 1 and Visit 2 and between Visit 2 and Visit 3.
12. Have ongoing or anticipated disability compensation or litigation issues, in the best judgment of the investigator.
13. Have a presence of any factors/conditions, medical or other, that in the judgment of the investigator may interfere with performance of study outcome measures, such as treatment-refractory history.
14. Have serious or unstable cardiovascular, hepatic, renal, metabolic, respiratory, or hematologic illness, symptomatic peripheral vascular disease, or other medical condition or psychiatric conditions that, in the opinion of investigator and study physician, would compromise participation or be likely to lead to hospitalization during the course of the study.
15. Are non-ambulatory or require the use of crutches or a walker.
16. Current suicidal or homicidal ideation necessitating clinical intervention or representing an imminent concern, or history of suicide attempt in the past 3 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-09-13 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C. Naylor, PhD, Principal Investigator — Durham VA Medical Center; Christine E Marx, MD, Study Director — Durham VA Medical Center
Locations (1):
- Durham VA Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Naylor JC, Kilts JD, Shampine LJ, Parke GJ, Wagner HR, Szabo ST, Smith KD, Allen TB, Telford-Marx EG, Dunn CE, Cuffe BT, O'Loughlin SH, Marx CE. Effect of Pregnenolone vs Placebo on Self-reported Chronic Low Back Pain Among US Military Veterans: A Randomized Clinical Trial. JAMA Netw Open. 2020 Mar 2;3(3):e200287. doi: 10.1001/jamanetworkopen.2020.0287. PMID 32119096

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregnenolone: Pregnenolone fixed escalating up to 500mg/day will consist of the following schedule:
  Visit 1 (week -1, screening visit) and pain symptom assessment (no study medication) Visit 2 (week 0) placebo lead-in (all participants) Visit 3 (week 1, baseline visit): 50mg PO, BID x 1 week, Visit 4 (week 2): 150mg PO, BID x 1 week, Visit 5 (week 3): 250mg PO, BID for two weeks. Visit 6 (week 5): No medication will be dispensed; study medication will be tapered by 100mg per day and then discontinued.
  Pregnenolone
- Placebo: Placebo will be administered exactly the same as the active comparator (pregnenolone) and will consist of the following schedule:
  Visit 1 (week -1, screening visit) and pain symptom assessment (no study medication) Visit 2 (week 0) placebo lead-in (all participants) Visit 3 (week 1, baseline visit): placebo PO, BID x 1 week, Visit 4 (week 2): placebo PO, BID x 1 week, Visit 5 (week 3): placebo PO, BID for two weeks. Visit 6 (week 5): No medication will be dispensed; study medication will be tapered in the exact manner as active study medication and then discontinued.
  Placebo
Period: Visit 3 (Randomization Visit)
Arm/Group | Pregnenolone | Placebo
Started | 45 | 49
Completed | 45 | 49
Not Completed | 0 | 0
Period: Visit 4
Arm/Group | Pregnenolone | Placebo
Started | 45 | 49
Completed | 45 | 48
Not Completed | 0 | 1
Period: Visit 5
Arm/Group | Pregnenolone | Placebo
Started | 45 | 48
Completed | 44 | 47
Not Completed | 1 | 1
Period: Visit 6
Arm/Group | Pregnenolone | Placebo
Started | 44 | 47
Completed | 41 | 42
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregnenolone | Placebo | Total
Number analyzed (Participants) | 45 | 49 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 49 | 94
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.48 (9.47) | 37.55 (10.25) | 37.52 (9.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 40 | 44 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 17 | 32
  White | 26 | 30 | 56
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 45 | 49 | 94

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity Rating (Visit 6-Baseline)
Description: Weekly mean of the 24-hour average pain severity scores recorded daily on an 11-point Likert scale, an ordinal scale ranging from 0 (no pain) to 10 (worst pain). The outcome measure is the change in scores before and after treatment. That is, the baseline and Visit 6 difference scores.
Time Frame: Difference Scores (Visit 6-Baseline)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 41 | 42
units on a scale | 4.11 (0.18) | 4.67 (0.17)
Statistical Analysis 1: Comparison: Pregnenolone vs Placebo; Test type: Superiority; p = 0.02, Mixed Models Analysis — a priori threshold set at 0.05; Mean Difference (Final Values) = -0.56, Standard Error of Mean 0.25

2. Secondary Outcome: Change in Pain Interference Scores (Visit 6-Baseline)
Description: The The Brief Pain Inventory (BPI) is a self-reported scale that measures the severity of pain and the interference of pain on function. The scores range from 0 (no pain) to 10 (pain as severe as you can imagine). There are 4 questions assessing worst pain, least pain, average pain in the past 24 hours, and the pain right now. The Interference scores range from 0 (does not interfere) to 10 (completely interferes). There are 7 questions assessing the interference of pain in the past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. The outcome measure is the change in scores before and after treatment. That is, the baseline and Visit 6 difference scores.
Time Frame: Difference Scores of Averaged Pain Interference Domains (Visit 6-Baseline)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 41 | 42
units on a scale | 1.84 (0.23) | 2.21 (0.26)
Statistical Analysis 1: Comparison: Pregnenolone vs Placebo; Test type: Superiority; p = 0.26, Mixed Models Analysis; Mean Difference (Final Values) = 0.83, Standard Error of Mean 0.14

3. Secondary Outcome: Change in Beck Depression Inventory (Visit 6-Baseline)
Description: The Beck Depression Inventory is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression (Beck, et al., 1961). Scores range from 0 (no depression) to 63 (severe depression). The outcome measure is the change in scores before and after treatment. That is, the baseline and Visit 6 difference scores.
Time Frame: Difference Scores of BDI (Visit 6-Baseline)
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 41 | 42
units on a scale | 6.06 (0.50) | 6.26 (0.66)
Statistical Analysis 1: Comparison: Pregnenolone vs Placebo; Test type: Superiority; p = 0.79, Mixed Models Analysis; Mean Difference (Final Values) = 0.97, Standard Error of Mean 0.12

4. Secondary Outcome: Change in Davidson Trauma Scale (Visit 6-Baseline)
Description: The Davidson Trauma Scale (DTS) is a 17-item self-report measure that assesses the 17 DSM-IV symptoms of PTSD. Items are rated on 5-point frequency (0 = "not at all" to 4 = "every day") and severity scales (0 = "not at all distressing" to 4 = "extremely distressing"). Respondents are asked to identify the trauma that is most disturbing to them and to rate, in the past week, how much trouble they have had with each symptom. The DTS yields a frequency score (ranging from 0 to 68), severity score (ranging from 0 to 68), and total score (ranging from 0 to 136). The outcome measure is the change in scores before and after treatment. That is, the baseline and Visit 6 difference scores.
Time Frame: Difference Scores of Total DTS Scores (Visit 6-Baseline)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 41 | 42
units on a scale | 17.71 (1.93) | 15.04 (11.70)
Statistical Analysis 1: Comparison: Pregnenolone vs Placebo; Test type: Superiority; p = 0.23, Mixed Models Analysis; Mean Difference (Final Values) = 1.18, Standard Error of Mean 0.16

5. Secondary Outcome: Change in Tower of London (Visit 6-Baseline)
Description: The Tower of London is a clinician administered subtest from the Brief Assessment of Cognition-Affect (BAC-A) which measures executive functioning. Participants were shown two pictures simultaneously. Each picture showed three balls of different colors arranged on three pegs, with the balls in a unique arrangement in each picture. Participants were asked to give the total number of times the balls in one picture need to be moved in order to make the arrangement of balls identical to that of the other, opposing picture. There were 20 trials, 2 more were added if all 10 prior trials were correct. Range of scores was 0-22, higher scores are better. Z scores calculated and reported. The outcome measure is the change in Z scores before and after treatment. That is, the baseline and Visit 6 difference scores.
Time Frame: Difference Z-Score (Visit 6-Baseline)
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 41 | 42
units on a scale | 0.71 (0.08) | 0.76 (0.07)
Statistical Analysis 1: Comparison: Pregnenolone vs Placebo; Test type: Superiority; p = 0.63, Mixed Models Analysis; Mean Difference (Final Values) = 0.93, Standard Error of Mean 0.13

6. Secondary Outcome: Change in Digit Sequence (Visit 6-Baseline)
Description: Digit Sequencing Task is a clinician administered subtest from the Brief Assessment of Cognition-Affect (BAC-A) which measures working memory and attention. Participants were presented with clusters of numbers of increasing length.They were asked to tell the experimenter the numbers in order, from lowest to highest. Measures: number of correct responses (range: 0-28, higher is better). Scores converted to Z-scores. The outcome measure is the change in Z scores before and after treatment. That is, the baseline and Visit 6 difference scores.
Time Frame: Difference Z-Scores (Visit 6-Baseline)
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 41 | 42
units on a scale | 0.79 (0.06) | 0.74 (0.07)
Statistical Analysis 1: Comparison: Pregnenolone vs Placebo; Test type: Superiority; p = 0.62, Mixed Models Analysis; Mean Difference (Final Values) = 1.06, Standard Error of Mean 0.13

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected at each visit throughout study participation and by phone two weeks post study completion, up to 8 weeks.
Groups:
- Pregnenolone: Pregnenolone fixed escalating up to 500mg/day with following schedule:
  Visit 1 (week -1, screening visit) and pain symptom assessment (no study medication) Visit 2 (week 0) placebo lead-in (all participants) Visit 3 (week 1, baseline visit): 50mg PO, BID x 1 week, Visit 4 (week 2): 150mg PO, BID x 1 week, Visit 5 (week 3): 250mg PO, BID for two weeks. Visit 6 (week 5): No medication will be dispensed; study medication will be tapered by 100mg per day and then discontinued.
  Pregnenolone
- Placebo: Placebo was administered exactly the same as the active comparator (pregnenolone) with the following schedule:
  Visit 1 (week -1, screening visit) and pain symptom assessment (no study medication) Visit 2 (week 0) placebo lead-in (all participants) Visit 3 (week 1, baseline visit): placebo PO, BID x 1 week, Visit 4 (week 2): placebo PO, BID x 1 week, Visit 5 (week 3): placebo PO, BID for two weeks. Visit 6 (week 5): No medication will be dispensed; study medication will be tapered in the exact manner as active study medication and then discontinued.
  Placebo
Arm/Group | Pregnenolone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/49
Other Adverse Events (participants affected / at risk) | 6/45 | 6/49
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregnenolone (N=45) | Placebo (N=49)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Decreased Appetite (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Drowsiness (General disorders) | 1 (1) | 1 (2)
Dry Mouth (General disorders) | 1 (2) | 2 (2)
Headache (General disorders) | 1 (2) | 2 (3)
Insomnia (General disorders) | 1 (4) | 0 (0)
Myoclonus (General disorders) | 0 (0) | 1 (1)
Nausea (General disorders) | 0 (0) | 1 (1)
Paresthesia (General disorders) | 0 (0) | 1 (1)
Tremor (General disorders) | 0 (0) | 1 (2)
Urinary Retention (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT01898013/Prot_SAP_000.pdf